CLINICAL TRIAL: NCT04123457
Title: Biorepository for Discovery and Validation of Biomarkers for Optimization of Microvascular Treatment of Lymphedema
Brief Title: Biorepository of Biomarkers for Optimization of Microvascular Treatment of Lymphedema
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Antonio J. Forte, Principal Investigator, Mayo Clinic
Other Study IDs: 18-006576
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers are collecting information, saliva, blood and tissue from subjects with lymphedema to store for future research.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Ability to provide written consent
* Has been diagnosed with Lymphedema

Exclusion Criteria:

* Under the age of 18 years old
* Inability to provide written consent
* Previous lymphovenous bypass or lymph node transfer surgery
* Major changes occur to co-morbid conditions
* Proven ICG or iodine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of Lymphedema.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Biospecimen Acquisition | 1 year
  Number of biospecimens collected

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Forte, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials